CLINICAL TRIAL: NCT05004038
Title: A Phase IIA Randomized Double-blind Placebo-controlled Single-centre Study of the Effect of Bacillus Calmette-Guérin (BCG) Vaccination on the HIV Latent Reservoir
Brief Title: BCG Vaccination Effect on Latent Reservoir Size in Treated HIV-1 Infection:
Acronym: BELIEVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-01481
Record Dates: First submitted 2021-07-12; First posted 2021-08-13 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: A phase IIA randomized double-blind placebo-controlled single-centre study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Group (Active Comparator): We will conduct a randomized, double-blind trial using a stepped-wedge design and involving a total of 60 patients with stable treated HIV and suppressed viral load who will all receive the BCG vaccine during the course of the study. Patients will be divided into two groups of equal size (early and late groups regarding administration of the BCG verum). The trial will be placebo-controlled and double-blind. Patients in the early group will receive the BCG verum at the beginning of Treatment Phase 1, and then the placebo at the beginning of Treatment Phase 2.
  Interventions: Biological: BCG Vaccine AJVaccines
- Late Group (Active Comparator): Patients in the late group will receive placebo at the beginning of Treatment Phase 1 and then the BCG verum at the beginning of Treatment Phase 2.
  Interventions: Biological: BCG Vaccine AJVaccines

INTERVENTIONS:
Biological: BCG Vaccine AJVaccines — Single intradermal injection of BCG Vaccine according to published Summary of Product Characteristics

SUMMARY:
A phase IIA randomized double-blind placebo-controlled single-centre study of the effect of Bacillus Calmette-Guérin (BCG) vaccination on the HIV latent reservoir

DETAILED DESCRIPTION:
Background and Rationale:

HIV infection affects around 40 million people globally and is incurable due to persistence of viral genetic material within the host genome as the latent reservoir. Patients within the Swiss HIV Cohort Study with latent tuberculosis were recently shown to have a reduced set point HIV viral load compared to tuberculosis (TB)-naïve individuals. The BCG vaccine has been shown to have wide-ranging immunostimulatory effects and can simulate latent tuberculosis infection.

Objective(s):

The purpose of this study is to characterise potential sustained and clinically relevant effects of the BCG vaccine on the size of the latent HIV-1 reservoir in individuals with stable treated HIV-1 infection with suppressed viremia.

The study seeks primarily to determine the effect of a single dose of the BCG vaccine on the size of the latent HIV-1 viral reservoir over a period of up to 6 months post-administration compared to the size at baseline.

Study design:

Monocentric, randomized, placebo-controlled, stepped-wedge study design with all patients receiving BCG either at baseline or after three months

Measurements and procedures:

Measurement of the HIV-1 latent reservoir using peripheral blood mononuclear cells at three monthly intervals beginning on Day 0.

Study Product / Intervention: Single intradermal application of BCG Vaccine AJVaccines powder for suspension for injection according to the manufacturers' instructions.

Control Intervention: Single intradermal application of 0.1ml of 0.9% saline placebo using an identical procedure.

Number of Participants with Rationale: The study involves 60 participants in total, divided equally between two groups, who will receive early or late administration of the BCG vaccine.

Study Duration: The estimated study duration is 15 months

Statistical Considerations:

In order to power the trial to detect a relevant reduction of the HIV-1 latent reservoir with 90% certainty with a power of 80% at a probability of type 1 error of 5%, we need to enrol 54 patients (based on a paired t-test power calculation assuming the effect size mentioned in Section 10 and the variance of log- total HIV-1 DNA observed by Bachmann et al1). Assuming a drop-out of 10% this implies that 60 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (see Informed Consent Form),
* Age ≥18 years,
* HIV-1 infection under continuous antiretroviral therapy for ≥1.5 years as requested in the Systems X Cohort,
* Current participation in the Swiss HIV Cohort Study and past participation in the Systems X Cohort.

Exclusion Criteria:

* History of virological failure or treatment interruption at any time, defined as HIV-1 viral load >200c/ml at two consecutive measurements at least 4 weeks apart,
* CD4 T-cell count <200/μl at any time or <350/μl during the past 1 year
* Presence of other relevant immunosuppression according to the investigator in addition to HIV (a daily steroid intake of ≥20mg is considered clinically relevant),
* History of or current clinical evidence of active tuberculosis,
* Previous positive tuberculin skin test or tuberculosis INF-gamma release assay (Quantiferon-Test) within the past 10 years,
* Previous BCG-vaccination within the past 10 years,
* Known allergy to BCG vaccine or any of its components,
* Documented current febrile illness at screening or in the past 7 days.
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in size of the HIV-1 latent reservoir at 6 months | 6 months for each patient
  The primary outcome will be the change in size of the HIV-1 latent reservoir at 6 months post-BCG vaccination compared to pre-vaccination in all patients, with each patient serving as their own control.
  This HIV-1 latent reservoir size will be measured as total HIV-1 DNA in peripheral blood mononuclear cells, a well-established and extensively validated marker for the HIV-1 reservoir found to be sensitive, clinically relevant and feasible in larger populations.

SECONDARY OUTCOMES:
The change in size of the HIV-1 latent reservoir at 3 months | 3 months for each patient
  The change in size of the HIV-1 latent reservoir at 3 months post-BCG vaccination compared to 3 months post-placebo (early group versus late group at day 90)
The change in size of the HIV-1 latent reservoir at 3 months (in all patients) and 9 months (in the early group) post-BCG vaccination compared to pre-vaccination | 9 months for each patient
  The change in size of the HIV-1 latent reservoir at 3 months (in all patients) and 9 months (in the early group) post-BCG vaccination compared to pre-vaccination
The frequency and incidence of adverse events of interest in the verum group compared to the placebo group | 9 months
  The frequency and incidence of adverse events of interest in the verum group compared to the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Nemeth, Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No